CLINICAL TRIAL: NCT01061281
Title: Evaluation of the Tecnis™ Multifocal and Crystalens™ Accommodating Intraocular Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Farrell Tyson, Cape Coral Eye Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tecnis MF/Crystalens
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Aphakia
Keywords: Aphakia following refractive lensectomy to treat presbyopia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecnis MF IOL (Active Comparator)
  Interventions: Device: Tecnis MF IOL
- Crystalens AO IOL (Active Comparator)
  Interventions: Device: Crystalens AO IOL

INTERVENTIONS:
Device: Tecnis MF IOL — 20 patients enrolled with the Tecnis MF IOL.
  Arms: Tecnis MF IOL
Device: Crystalens AO IOL — 20 patients enrolled with the Crystalens AO
  Arms: Crystalens AO IOL

SUMMARY:
The purpose of this study is to compare the visual outcomes with bilateral implantation of Tecnis MF and Crystalens™ AO Aberration-free Accommodating intraocular lens (IOLs) 6 months after post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation has been planned for both eyes
* Visual potential of 20/25 or better in each eye after cataract removal and IOL implantation
* Preoperative best-corrected distance visual acuity (BCDVA) worse than 20/40 Snellen
* Naturally dilated pupil size (in dim light) > 4.0 mm (with no dilation medications) for both eyes
* Preoperative corneal astigmatism of 1.0 D or less
* Clear intraocular media other than cataract
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Subjects with diabetes mellitus
* Uncontrolled systemic or ocular disease
* History of ocular trauma or prior ocular surgery
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Contact lens usage within 6 months for PMMA contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lenses
* Requiring an intraocular lens < 15.0 or > 26.0 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Refraction | 1 year
Distance Visual Acuities | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Farrell Tyson, Cape Coral, Florida, United States